CLINICAL TRIAL: NCT00489931
Title: A Phase I Open-Label Study of the Safety and Immunogenicity of a Recombinant DNA Plasmid Vaccine, VRC-AVIDNA036-00-VP, Encoding for the Influenza Virus H5 Hemagglutinin Protein Administered Intradermally in Healthy Adults
Brief Title: Phase I Open-Label Study of Recombinant DNA Plasmid Vaccine, VRC-AVIDNA036-00-VP, Encoding for Influenza Virus H5 Hemagglutinin Protein Given Intradermally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 070172; 07-I-0172
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-15

CONDITIONS: Influenza A Virus, H5N1 Subtype; Influenza A Virus; Influenzavirus A; Orthomyxovirdae; H5N1 Virus
Keywords: Avian Influenza; Healthy; Immunity; Preventive; Bird Flu; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza in Birds

INTERVENTIONS:
Drug: VRC-AVIDNA036-00-VP

SUMMARY:
This study will evaluate the safety and effectiveness of a vaccine to prevent avian influenza (bird flu). About 25 to 50 million cases of influenza occur a year in the U.S., leading to 150,000 hospitalizations and 30,000 to 40,000 deaths. Globally, a pandemic influenza may be 1 billion flu cases, with 3 to 5 million cases of severe illness and up to half a million deaths annually. There is potential threat of a pandemic from emerging virus strains for which the population has little or no preexisting immunity. Avian influenza A (H5N1) viruses causing serious disease have emerged recently, affecting domestic and wild bird populations.

Patients ages 18 to 60 who are in good health and not pregnant or breast feeding may be eligible for this study. The study will be done at the NIH Clinical Center by staff of the Vaccine Research Center. It will last about 32 weeks for each person. A traditional needle or a needle-free device called Biojector 2000 will be used. Intramuscular (in the muscle) and subcutaneous (in fat below the skin) delivery of vaccine via Biojector is cleared for use by the Food and Drug Administration and is not considered investigational. Intradermal (in the skin) delivery of vaccine by Biojector in this study is deemed investigational but has been evaluated in humans before, and found safe and well tolerated in other trials.

There will be about 10 clinic visits in this study, and it is important to stay on schedule. Visits are about 2 hours, though on injection days, visits are about 4 hours. Injections are given on day 0 and at weeks 4 and 8. The vaccine is given by injections in the skin on the upper arms. Clinic staff will observe patients for 30 minutes after each vaccination. One to 2 days after the first injection, there will be a clinic visit. One to 3 days after the second and third injections, patients need to telephone clinic staff to report on how they are doing. Patients will complete a diary card at home, recording temperature and symptoms, and looking at the injection site daily for 5 days. Patients should report any side effects to one of the study physicians or nurses as soon as possible. They will return to the clinic 2 weeks after each injection. A needle-free system uses the pressure of carbon dioxide, instead of a needle, to inject the vaccine into the skin. Discomfort can result from either the needle-free device or the needle. There may be stinging, pain, soreness, swelling, bruising, or a small cut in the skin.

DETAILED DESCRIPTION:
Study Design: This is a Phase I study to evaluate safety, tolerability, and immunogenicity of a recombinant DNA vaccine against the influenza virus H5 hemagglutinin by intradermal (ID) delivery. The hypothesis is that this vaccine will be safe for human administration by ID delivery by either needle/syringe or Biojector and will elicit antibody and T cell responses against the H5 protein. Primary objectives are to evaluate safety and tolerability of the vaccine at 500 micrograms ID administered by needle and syringe or by Biojector and at 1 mg ID administered by Biojector as two injections in the same or in different arms in healthy adults. Secondary and exploratory objectives are related to immunogenicity.

Product Description: The vaccine is composed of a single closed-circular DNA plasmid that encodes the H5 protein with a CMV/R promoter. Vaccine vials will be supplied at 4 mg/mL. Each injection will be 125 microliters (500 micrograms) administered ID over the deltoid muscle using the Biojector® (Registered Trademark) 2000 Needle-Free Injection Management System (Biojector) or needle and syringe.

Subjects: A total of 40 healthy adults, ages 18-60 years will be enrolled.

Study Plan: Subjects will be simultaneously randomized at a ratio of 1:1:1:1 into one of four groups as shown in the schema. The protocol requires ten clinic visits and three telephone follow-up contacts.

Study Duration: Each participant will complete 32 weeks of clinical follow up.

Study Endpoints: The primary endpoint is safety and tolerability of the regimen. The secondary immunogenicity endpoint is H5-specific antibody as measured by hemagglutination inhibition (HAI) assay and H5 neutralizing antibody assay at Study Week 12. Other immunogenicity assays at timepoints throughout the study may also be completed as exploratory evaluations.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 60 years old.
2. Available for clinical follow-up through Week 32.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to donate blood for sample storage to be used for future research.
7. In good general health without clinically significant medical history.
8. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than 40 within the 28 days prior to enrollment.

   Laboratory Criteria within 28 days prior to enrollment:
9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
10. White blood cells (WBC) = 3,300-12,000 cells/mm(3)
11. Differential either within institutional normal range or accompanied by site physician approval
12. Total lymphocyte count greater than or equal to 800 cells/mm(3)
13. Platelets = 125,000 - 500,000/mm(3)
14. Alanine aminotransferase (ALT) less than or equal to 1.25 upper limit of normal
15. Serum creatinine less than or equal to 1 times upper limit of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males)
16. Normal urinalysis, defined as negative glucose, negative or trace protein and no clinically significant blood in the urine.
17. Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study]
18. Negative hepatitis B surface antigen (HBsAg)
19. Negative anti-hepatitis C virus (HCV) antibody and negative HCV PCR.
20. Negative for active elicit drug abuse for amphetamines, barbiturates, cocaine, lysergic acid diethylamine (LSD), opiates, or phencyclidine, based on history and urine drug screen performed at the NIH Clinical Center.

    Female-Specific Criteria:
21. Negative beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential (i.e., women who have had surgical hysterectomy will not require pregnancy testing).
22. A female participant must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 26 of the study,

OR

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 26 of the study by one of the following methods: condoms, male or female, with or without a spermicide; diaphragm or cervical cap with spermicide; intrauterine device; contraceptive pills, patch, implant or any other FDA-approved contraceptive method; male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply.

Women Specific:

1. Breast-feeding or planning to become pregnant during the study.

   Volunteer has received any of the following substances:
2. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past three months.

   [Note: The following will NOT exclude study participation:

   use of corticosteroid nasal spray for rhinitis

   topical corticosteroids for an acute uncomplicated dermatitis

   short-acting beta-agonists in controlled asthmatics

   a short course (10 days or less) of corticosteroids for a non-chronic condition completed at least 2 weeks prior to enrollment in this study]
3. Blood products within 120 days prior to HIV screening
4. Immunoglobulin within 60 days prior to HIV screening
5. Live attenuated vaccines within 30 days prior to initial study vaccine administration
6. Investigational research agents within 30 days prior to initial study vaccine administration
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration
8. Current anti-TB prophylaxis or therapy
9. Previous H5 avian influenza investigational vaccine.

   Volunteer has a history of any of the following clinically significant conditions:
10. Autoimmune disease or immunodeficiency.
11. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
12. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
13. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
15. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
16. Idiopathic urticaria within the past 2 years
17. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
18. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with injections or blood draws.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Allergic reaction to aminoglycoside antibiotics.
23. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, a history of suicide plan or attempt.
24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44
Dates: Start 2007-06-18; Study Completion 2009-04-15

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Taubenberger JK, Reid AH, Lourens RM, Wang R, Jin G, Fanning TG. Characterization of the 1918 influenza virus polymerase genes. Nature. 2005 Oct 6;437(7060):889-93. doi: 10.1038/nature04230. PMID 16208372